CLINICAL TRIAL: NCT01719302
Title: Phase I/II Study of the Combination of Docetaxel, Gemcitabine and Pazopanib for Neoadjuvant Treatment of Patients With Operable Soft Tissue Sarcoma
Brief Title: Docetaxel, Gemcitabine and Pazopanib as Treatment for Soft Tissue Sarcoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Claire Verschraegen, Director, Hematology Oncology Unit, University of Vermont
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VCC 1202
Record Dates: First submitted 2012-10-29; First posted 2012-11-01 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Stage III Adult Soft Tissue Sarcoma
Keywords: Soft tissue sarcoma; gemcitabine; docetaxel; pazopanib
MeSH Terms: conditions — Sarcoma | interventions — Gemcitabine; Docetaxel; pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cohort 1 (Experimental)
  Interventions: Drug: Gemcitabine; Drug: Docetaxel; Drug: Pazopanib

INTERVENTIONS:
Drug: Gemcitabine — 1500 mg/m^2 given days 1 and 15 of every 28 day cycle for a total of 4 cycles
  Other Names: Gemzar
Drug: Docetaxel — 50 mg/m^2 on days 1 and 15 of each 28 day cycle for a total of 4 cycles
  Other Names: Taxotere
Drug: Pazopanib — Starting dose of 400 mg/day starting 72 hours after docetaxel/gemcitabine administration for 10 days (days 4-13 and 18-27) of each 28 day cycle for a total of 4 cycles. Dose will be increased by 200 mg/day for each cohort until the maximum tolerated dose is identified.
  Other Names: Votrient

SUMMARY:
Chemotherapy treatment with docetaxel and gemcitabine is a standard treatment for patients with soft tissue sarcoma. This study is designed to explore whether the addition of tyrosine kinase inhibitor pazopanib enhances the anticancer effect of the chemotherapy drugs.

The Phase I component of this study is designed to determine the maximum tolerated dose of pazopanib when given with docetaxel and gemcitabine. The Phase II component is designed to determine the overall response rate of the combination of docetaxel, gemcitabine and pazopanib prior to surgical resection in patients with soft tissue sarcoma.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* chemotherapy naive, histologically high grade soft tissue sarcoma that is considered to be operable
* tumor greater than 5 cm in longest dimension
* life expectancy of at least 6 months
* Zubrod performance status of 0-2
* signed informed consent
* adequate bone marrow function defined by:

  1. absolute peripheral granulocyte count of >1500 cells/mm^3
  2. hemoglobin >8.0 g/dl
  3. platelet count >100,000/mm^3
  4. absence of a regular red blood cell transfusion requirement
* adequate hepatic function defined by:

  1. total bilirubin <1.5 x upper limit of normal (ULN)
  2. AST, ALT and alkaline phosphatase all not more than 2.5 x ULN
* adequate renal function defined by:

  1. serum creatinine <1.5 x ULN
* negative pregnancy test for women of child bearing potential
* willingness to use effective contraception while on treatment and for 3 months thereafter

Exclusion Criteria:

* Multiple metastases (patients with 5 or fewer oligometastases that could be resectable are eligible)
* Pregnant women or nursing mothers
* concurrent chemotherapy or radiation therapy
* severe medical problems (at the discretion of the investigator)
* history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80
* symptomatic brain metastases
* cirrhosis
* dermatofibrosarcoma protuberans (DFSP), embryonal rhabdomyosarcoma or alveolar soft part sarcoma (ASPS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 1 cycle (28 days)

SECONDARY OUTCOMES:
Overall response rate | 4 cycles (112 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Fletcher Allen Health Care, Burlington, Vermont, United States